CLINICAL TRIAL: NCT02049788
Title: Effects of a Low Glycemic Index Diet on Body Composition and Metabolic Syndrome Risks in Obese Thai Children: A Randomized Controlled Trial
Brief Title: Effects of a Low Glycemic Index in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGI-01
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low calorie/fat diet (Active Comparator): The low calorie/fat diet group, obese children aged 9-16, received conventional behavioural lifestyle modification instructions x 1/month for 6 months about low-calorie (approximately 1200-1300 kcal/day), low-fat (25% of total calories from fat) and about physical activity (increase non-weight bearing exercise 30 minutes/day at least x 3 times/week, increase physical activity in their routine and decrease sedentary activity).
  Interventions: Behavioral: low calorie/fat diet
- Low glycaemic index diet (Experimental): Low glycaemic index diet group, obese children of both sexes aged 9-16, received experimental behavioural lifestyle modification instructions x 1/month for 6 months about low glycaemic index diet (selection of low-GI carbohydrates with the caloric distribution of carbohydrate 50-55%: protein 15-20%: fat 30-35%, instruction by two-hour small classes with parental participation low GI cooking demonstration and food labeling guidance) and about physical activity (increase non-weight bearing exercise 30 minutes/day at least x 3/week, increase physical activity in their routine and decrease sedentary activity).
  Interventions: Behavioral: Low glycaemic index diet

INTERVENTIONS:
Behavioral: low calorie/fat diet — Conventional behavioural lifestyle modification instructions x 1/month for 6 months about low-calorie (approximately 1200-1300 kcal/day), low-fat (25% of total calories from fat) and about physical activity (increase non-weight bearing exercise 30 minutes/day at least x 3 times/week, increase physical activity in their routine and decrease sedentary activity).
  Arms: low calorie/fat diet
Behavioral: Low glycaemic index diet — Experimental behavioural lifestyle modification instructions x 1/month for 6 months about low glycaemic index diet (selection of low-GI carbohydrates with the caloric distribution of carbohydrate 50-55%: protein 15-20%: fat 30-35%, instruction by two-hour small classes with parental participation low GI cooking demonstration and food labeling guidance) and about physical activity (increase non-weight bearing exercise 30 minutes/day at least x 3/week, increase physical activity in their routine and decrease sedentary activity).
  Arms: Low glycaemic index diet

SUMMARY:
The objective of this study is to compare the effectiveness of a low-GI diet program and a standard counseling program in the treatment of obese Thai children.

DETAILED DESCRIPTION:
Obese children aged 9-16 years from King Chulalongkorn Memorial Hospital were randomized to receive instruction either for a low-GI diet (intervention group) or a low-calorie, low-fat diet (control group). Both groups were followed-up every month for six months. The primary outcomes were body composition changes during the six-month period, measured by dual X-ray absorptiometry (DEXA) and bioelectrical impedance analysis (BIA). Secondary outcomes were metabolic syndrome risk changes measured by fasting plasma glucose, insulin, and lipid profiles.

The adherence to the nutritional education and physical activity recommendation was evaluated by using three-day dietary records (two weekdays and one weekend day) and a physical activity questionnaire at each visit. All participants were examined and counseled about physical activity and life style modification strategies by a pediatrician at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between nine to sixteen years old
* BMI higher than the International Obesity Task Force cut-off

Exclusion Criteria:

* psychological problems
* underlying diseases that might affect a weight management program
* used drugs associated with weight increment or reduction
* attended other weight management programs

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition measured by BIA and DEXA at month 6 | 6 months

SECONDARY OUTCOMES:
Change from baseline in metabolic syndrome risks at month 6 | 6 months
  Metabolic syndrome risks are fasting blood sugar, insulin and lipid profiles.

OTHER OUTCOMES:
Change from baseline in body weight, BMI z-score and waist circumference at month 6 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sirinuch Chomtho, M.D., PhD., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Patumwan, Bangkok, Thailand